CLINICAL TRIAL: NCT01279382
Title: Effectiviteit Van Hypnotherapie Bij Prikkelbare Darmsyndroom (Effectiveness of Hypnotherapy in Irritable Bowel Syndrome)
Brief Title: Effect of Hypnotherapy in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. Dr. A. Masclee, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P113/99
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Symptoms; Psychological status; Hypnotherapy; Relaxation training
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Hypnosis; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Care as usual (CON) (Other): CON was given to a subgroup of patients as control treatment in IBS treatment
  Interventions: Other: Care as usual (CON)
- Hypnotherapy (HYP) (Other): HYP was given to a subgroup of patients as intervention in IBS treatment
  Interventions: Behavioral: Hypnotherapy (HYP)
- Relaxation training (RT) (Other): RT was given to a subgroup of patients as intervention in IBS treatment
  Interventions: Behavioral: Relaxation training (RT)

INTERVENTIONS:
Behavioral: Hypnotherapy (HYP) — Hypnotherapy was given to a subgroup of patients as intervention in IBS treatment
  Arms: Hypnotherapy (HYP)
Behavioral: Relaxation training (RT) — RT was given to a subgroup of patients as intervention in IBS treatment
  Arms: Relaxation training (RT)
Other: Care as usual (CON) — CON was given to a subgroup of patients as control intervention in IBS treatment
  Arms: Care as usual (CON)

SUMMARY:
In this trial, the effects of two psychological interventions - i.e. hypnotherapy and relaxation training - are compared with care as usual in IBS treatment. The investigators hypothesized that hypnotherapy is most effective in reducing complaints in IBS.

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome (Rome II)
* Presence of complaints < 12 months

Exclusion Criteria:

* Gastrointestinal disorders, other than IBS
* Previous psychotherapeutic treatment for IBS
* Severe psychological comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-01; Study Completion 2006-01

PRIMARY OUTCOMES:
Mean symptom score (MSS)

SECONDARY OUTCOMES:
Psychological measures, i.e. anxiety and depression (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, Prof. Dr., Principal Investigator — Head of dept
Locations (1):
- LUMC - Leiden, Leiden, Netherlands